CLINICAL TRIAL: NCT00964639
Title: Postoperative Pain in Children With Cerebral Palsy After Pelvic and Femoral Osteotomies. A Prospective, Randomized and Double-blinded Study
Brief Title: Postoperative Pain in Children With Cerebral Palsy After Pelvic and Femoral Osteotomies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FLACC2008
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Postoperative Pain; Cerebral Palsy
Keywords: Pain; Postoperative; Local infiltration analgesia; Cerebral palsy; r-FLACC
MeSH Terms: conditions — Pain, Postoperative; Cerebral Palsy; Pain | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline (Placebo Comparator)
  Interventions: Drug: Saline
- Naropin (Active Comparator)
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — During the surgery infiltration with Naropine 2 mg/ml. The dosage in the infiltration is 2 mg/kg. Thereafter bolus 3 times a day
  Arms: Naropin
Drug: Saline — During the surgery infiltration with saline. Thereafter bolus 3 times a day
  Arms: Saline

SUMMARY:
This study is a comparison of postoperative pain in children with cerebral palsy after surgery on the hip or femur. One group is treated with p.o. (by mouth) or intravenous (i.v.) analgesia, and the other group is treated with local infiltration analgesia with Naropine.

Pain is measured with r-FLACC, a pain-score validated for children with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Age under 18
* informed consent
* Postoperative cast with spica

Exclusion Criteria:

* Previous surgery in the same hip
* Other surgical procedure planned at the same time
* Bilateral surgery
* Previous allergic reaction to local analgesia

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2009-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Difference in pain measured with r-FLACC between the 2 groups | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Departement of childrens orthopaedics, Aarhus University Hospital, Aarhus, Denmark